CLINICAL TRIAL: NCT05426837
Title: Combating Social Isolation in Older Adults: Randomized Clinical Trial Evaluating the Acceptability and Efficacy of a Brief, Technology Delivered Intervention
Brief Title: Combatting Social Isolation in Older Adults
Acronym: CSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Retirement Research Foundation (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Distinguished Research Professor, Florida State University
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003135
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-11

CONDITIONS: Loneliness; Social Isolation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: Following the production of the refined/modified CSI, a RCT will be initiated to assess the efficacy of the CSI intervention relative to a Health Education Training (HET) control group.
  Approximately 50 participants will be randomly assigned to one of two conditions (1) CSI or (2) HET Control. Consistent with the rationale of an Indicated clinical trial, the primary entry criteria will be age (>65) as well as above average levels of loneliness (primary outcome). Participants will be assessed on a range of relevant outcome measures at pretreatment, post-treatment, and 1-month follow-ups. There are three interrelated study hypotheses (see Aim 2 above):
  1. CSI will significantly reduce loneliness relative to control.
  2. CSI will positively impact other outcomes such as quality of life during the follow-up period relative to control.
  3. Intervention related changes in risk (PB/TB) will mediate the relationship between CSI and outcomes (loneliness) at follow-up.
Who Masked: Participant
Masking Description: Participants will be randomized to receive either control or intervention condition and they will be blind to which condition they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health Education Training (Placebo Comparator): Health Education Training (HET) control condition covers standard healthy lifestyle behaviors as well as broad coping strategies to address stress. HET is a fully computerized 1-hour control condition focused on increasing healthy behaviors and decreasing unhealthy behaviors. Content includes healthy eating, hydration, sleep and rest, exercise, stress management as well as other healthy lifestyle tips. The HET protocol has been used in prior studies as a control condition for CSI to account for intervention modality and time (e.g. Schmidt et al., 2014). HET is perceived positively, with high rates of acceptability. Importantly, HET is inert with respect to the proposed mechanism of action (PB/TB) (Schmidt et al., 2014; Schmidt et al., 2007; Short et al., 2015). Also, home practice will be prescribed to match the procedures used in CSI and practice forms are provided wherein participants will self-monitor some of the behaviors addressed in HET.
  Interventions: Behavioral: Health Education Training
- Combatting Social Isolation (Active Comparator): Combating Social Isolation (CSI). CSI and a similar version of this intervention called "Building Stronger Allies", has gone through a rigorous treatment development phase, pilot RCT, and larger RCTs (Schmidt et al., 2014; Schmidt et al., 2017; Schmidt et al., 2007; Norr et al., 2017; Short et al., 2015; Short et al., 2017a; Schmidt et al., submitted for publication). CSI is a transdiagnostic cognitive behavioral therapy (CBT)-based protocol designed to address elevated perceived burdensomeness (PB) and thwarted belongingness (TB). The CSI intervention was designed in consultation with clinicians experienced in treating individuals dealing with issues related to PB/TB. CSI is a fully computerized, 1-hour intervention. The latest version of CSI uses Vyond software for video animation and audio narration throughout, as well as interactive features (e.g., brief quizzes to promote comprehension). Procedures draw heavily on standard CBT techniques.
  Interventions: Behavioral: Combatting Social Isolation

INTERVENTIONS:
Behavioral: Combatting Social Isolation — A brief, computerized psychoeducational intervention designed to target ways to cope with and address loneliness and social isolation in older adults modeled after our group's previous Building Stronger Allies (BSA) intervention.
  Arms: Combatting Social Isolation
Behavioral: Health Education Training — Control condition where participants learn about healthy lifestyle behaviors.
  Other Names: Control
  Arms: Health Education Training

SUMMARY:
Increasing evidence suggests that perceived social isolation and loneliness are major risk factors for physical and mental illness in later life. The prevalence of loneliness in US older adults warrants concern, with an estimated 30% of American adults aged 70 years and older reporting heightened loneliness. A wide variety of interventions have been developed to address social isolation and loneliness ranging from social facilitation to animal therapies. While many intervention studies have attempted to address loneliness, social isolation and related constructs in older adults, this literature is underdeveloped and there is not an established or widely accepted set of treatments. Moreover, existing treatments tend to be lengthy, burdensome, and result in high dropout rates.

Brief, mechanism focused interventions are an alternative to more traditional forms of treatment. Because they are structured and brief, these treatments can be readily placed on the internet, making them extremely efficient, destigmatizing, and highly scalable. The investigators have developed and tested a web-based intervention called "Combating Social Isolation" (CSI) that the investigators believe offers an alternative to existing interventions for loneliness and social isolation in older adults. CSI evolved out of Interpersonal Theories of mood psychopathology (Joiner, 2005) and targets two risk factors central to social disconnection: perceived burdensomeness and thwarted belongingness (PB/TB). The investigators have one randomized clinical trial using CSI and are nearing completion of two other RCTs using this intervention. Evidence shows that CSI has very high levels of acceptability, and despite the brevity of the protocol (approximately 1 hour) can markedly impact loneliness. Moreover, reductions in these risk factors mediate later improvements in mental health outcomes and social disruption. The purpose of the current proposal is to adapt our existing protocol for older adults reporting loneliness and then obtain preliminary acceptability and efficacy data from a Phase II randomized clinical trial.

DETAILED DESCRIPTION:
The study design involves protocol refinement and clinical trial evaluation phases:

1. Refinement. The first phase of this proposal involves refining our existing protocol - "Combating Social Isolation" based on feedback from the target population (i.e., older adults experiencing loneliness). A small but representative sample of older adults (> age 64) (diversified by race, gender, and SES) from the Tallahassee metropolitan area will review the intervention and provide feedback (N approximately 12). The existing protocol includes psychoeducation about healthy relationships, "myth busting" around cognitive errors associated with loneliness (largely focused on social interaction) as well as skill building for social relationships. During the refinement phase, input from our collaborator with expertise in the development and use of technologies in older adults (Dr. Boot) will be utilized in an attempt to ensure good acceptability across the sample. Input from our collaborators specializing in interventions for older adults (Drs. Sheffler and Van Orden) will also be incorporated prior to and following feedback from participants. Feedback regarding ease of use, comprehension, limitations, and suggestions will be solicited using semi-structured interviews. Based on these assessments, the treatment will be redesigned accordingly. This phase is expected to take approximately 2 months. Note that the investigators have completed similar refinements for this intervention as well as others for particular populations (e.g., active duty military, first responders, Latinx) including the translation to different cultures and countries (e.g., Mexico, Japan, Germany, Australia).
2. Randomized Clinical Trial (RCT). Following refinement, the investigators will initiate a RCT focused on indicated prevention of adverse sequelae resulting from elevated loneliness. The final phase of the proposal will be used to determine the relative efficacy of the refined intervention versus a health education control condition. The rationale for an indicated prevention RCT is that only a subset of older adults' experiences significant loneliness. The investigators believe that this is an optimal target for an initial clinical trial for this intervention. An alternative approach would be to conduct a universal prevention RCT using a nonselected group of older adults. While the investigators believe that many (perhaps most) individuals would benefit from the information and skills covered in CSI, a more focused clinical trial at this stage would offer a more efficient means of demonstrating efficacy in the subgroup of older adults most likely to benefit from this intervention. Outcomes will be compared at post-treatment and at a one-month follow-up. The main dependent variables of interest will include loneliness, quality of interpersonal relationships and internalizing symptoms (anxiety and depression). This phase is expected to last 10 months.

Design Considerations. As with any project, there are a broad array of design options that may yield relevant information. In this section, the investigators summarize some of the key issues that contributed to the proposed study design.

Protocol Modification. Given that the existing protocol shows efficacy, there is some risk in modifying it. Therefore, our approach will be similar to other refinement studies where the investigators keep the core skills covered but substitute specific content areas with more relevant information. As noted above, the unique features of aging relevant to loneliness need to be incorporated (e.g., death of spouse, close friends, loss of independence). For example, one version of CSI includes vignettes and descriptions of active duty soldiers and Veterans that are unlikely to be relevant to many older adults. This content would be removed and replaced with vignettes featuring older adults with content that is appropriate and more typical for older adults.

Using a Semi-active Control Condition in the RCT. There are many different RCT designs that could be utilized including a waitlist control, which is likely to yield a larger effect size difference with the active intervention. However, prior studies suggest that CSI can outperform the proposed control condition, and this control condition helps to account for many confounds that a waitlist does not. Therefore, the investigators believe our choice of a stronger control group is warranted. Our "Healthy Lifestyle" control condition is also a web-based protocol that covers information and skills that many people believe to be helpful. Moreover, most participants find this control condition to be useful.

Limited Follow-up. Having a follow-up is important to demonstrate the initiation as well as some durability of treatment effects since the investigators would not expect immediate (post treatment) change in the outcomes of interest. As with any skill building protocol, time is needed for skills to be implemented. On the other hand, the duration of the grant period (12 months) limits the length of a viable follow-up period. The investigators believe that a one-month follow-up will be sufficient to show whether there are any treatment effects. Additional studies will be needed to demonstrate longer term benefits of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Access to text message reminders
* Elevated loneliness (i.e. higher than a score of 5 on the Hughes et al., 2004, Short Scale for Measuring Loneliness in Large Surveys)
* Treatment stability will be required in terms of both psychopharmacology (2 month stable dose) as well as psychotherapy (2 months of ongoing treatment).

Exclusion Criteria:

* Evidence of significant medical conditions including visual, auditory or cognitive impairments that would prevent comprehension of the intervention materials.
* Participants who change medications or initiate psychotherapy during the follow-up interval will be evaluated separately and potentially excluded from the main analyses.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
University of California Los Angeles Loneliness Scale | 1-month
  Scores range from 20-80 with higher scores indicating higher levels of loneliness.
Interpersonal Needs Questionnaire | 1-month
  Measures Perceived Burdensomeness & Thwarted belongingness - Scores from Thwarted Belongingness range from 9-63 with higher scores indicating more thwarted belongingness. Perceived burdensomeness scores range from 6-42 with higher scores indicating more perceived burdensomeness

SECONDARY OUTCOMES:
Berkman Social Network Inventory | 1-month
  Measures Structural Social Isolation with scores ranging from 0-infinity (scores are total number of people in their social network) and density of social network calculated depending on size of social network.
Patient Reported Outcomes Measurement Information System - Anxiety Short Form | 1-month
  Scores range from 8-40 with higher scores indicating more anxiety symptoms.
Patient Reported Outcomes Measurement Information System - Emotional Distress-Depression-Short Form | 1-month
  Scores range from 8-40 with higher scores indicating more depressive symptoms.
World Health Organization Quality of Life Scale (WHOQOL-Brief) | 1-month
  Scores range from 26-105 with higher scores indicating higher perceived quality of life.
Patient Reported Outcomes Measurement Information system - Perceived Stress | 1-month
  Scores range from 10-50 with higher scores indicating higher levels of perceived stress

OTHER OUTCOMES:
Schmidt Lab Acceptability Questionnaire | 1-month
  Semi-structured interviews will gauge participant attitudes toward the acceptability of and their satisfaction with with the CSI intervention. Scored items will range from 0-4 with higher scores indicating higher satisfaction with the intervention (e.g. how would you rate the quality of the intervention 0 being very low quality and 4 being very high quality).

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Schmidt, Ph.D, Principal Investigator — Florida State University
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers

REFERENCES:
- [Background] Berkman LF, Glass T, Brissette I, Seeman TE. From social integration to health: Durkheim in the new millennium. Soc Sci Med. 2000 Sep;51(6):843-57. doi: 10.1016/s0277-9536(00)00065-4. PMID 10972429
- [Background] Beland F, Zunzunegui MV, Alvarado B, Otero A, Del Ser T. Trajectories of cognitive decline and social relations. J Gerontol B Psychol Sci Soc Sci. 2005 Nov;60(6):P320-P330. doi: 10.1093/geronb/60.6.p320. PMID 16260706
- [Background] Aylaz R, Akturk U, Erci B, Ozturk H, Aslan H. Relationship between depression and loneliness in elderly and examination of influential factors. Arch Gerontol Geriatr. 2012 Nov-Dec;55(3):548-54. doi: 10.1016/j.archger.2012.03.006. Epub 2012 Apr 8. PMID 22487148
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Brummett BH, Barefoot JC, Siegler IC, Clapp-Channing NE, Lytle BL, Bosworth HB, Williams RB Jr, Mark DB. Characteristics of socially isolated patients with coronary artery disease who are at elevated risk for mortality. Psychosom Med. 2001 Mar-Apr;63(2):267-72. doi: 10.1097/00006842-200103000-00010. PMID 11292274
- [Background] Cacioppo JT, Hawkley LC, Crawford LE, Ernst JM, Burleson MH, Kowalewski RB, Malarkey WB, Van Cauter E, Berntson GG. Loneliness and health: potential mechanisms. Psychosom Med. 2002 May-Jun;64(3):407-17. doi: 10.1097/00006842-200205000-00005. PMID 12021415
- [Background] Cacioppo JT, Hawkley LC. Social isolation and health, with an emphasis on underlying mechanisms. Perspect Biol Med. 2003 Summer;46(3 Suppl):S39-52. PMID 14563073
- [Background] Cacioppo JT, Hughes ME, Waite LJ, Hawkley LC, Thisted RA. Loneliness as a specific risk factor for depressive symptoms: cross-sectional and longitudinal analyses. Psychol Aging. 2006 Mar;21(1):140-51. doi: 10.1037/0882-7974.21.1.140. PMID 16594799
- [Background] Cacioppo S, Grippo AJ, London S, Goossens L, Cacioppo JT. Loneliness: clinical import and interventions. Perspect Psychol Sci. 2015 Mar;10(2):238-49. doi: 10.1177/1745691615570616. PMID 25866548
- [Background] Sander R. Preventing social isolation and loneliness among older people: a systematic review of health promotion interventions. Nurs Older People. 2005 Mar 1;17(1):40. doi: 10.7748/nop.17.1.40.s11. PMID 27736564
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] Cohen S, Doyle WJ, Skoner DP, Rabin BS, Gwaltney JM Jr. Social ties and susceptibility to the common cold. JAMA. 1997 Jun 25;277(24):1940-4. PMID 9200634
- [Background] Cohen-Mansfield J, Perach R. Interventions for alleviating loneliness among older persons: a critical review. Am J Health Promot. 2015 Jan-Feb;29(3):e109-25. doi: 10.4278/ajhp.130418-LIT-182. PMID 24575725
- [Background] Cornwell EY, Waite LJ. Measuring social isolation among older adults using multiple indicators from the NSHAP study. J Gerontol B Psychol Sci Soc Sci. 2009 Nov;64 Suppl 1(Suppl 1):i38-46. doi: 10.1093/geronb/gbp037. Epub 2009 Jun 9. PMID 19508982
- [Background] Eng PM, Rimm EB, Fitzmaurice G, Kawachi I. Social ties and change in social ties in relation to subsequent total and cause-specific mortality and coronary heart disease incidence in men. Am J Epidemiol. 2002 Apr 15;155(8):700-9. doi: 10.1093/aje/155.8.700. PMID 11943687
- [Background] Dickens AP, Richards SH, Greaves CJ, Campbell JL. Interventions targeting social isolation in older people: a systematic review. BMC Public Health. 2011 Aug 15;11:647. doi: 10.1186/1471-2458-11-647. PMID 21843337
- [Background] Chastin S, Gardiner PA, Harvey JA, Leask CF, Jerez-Roig J, Rosenberg D, Ashe MC, Helbostad JL, Skelton DA. Interventions for reducing sedentary behaviour in community-dwelling older adults. Cochrane Database Syst Rev. 2021 Jun 25;6(6):CD012784. doi: 10.1002/14651858.CD012784.pub2. PMID 34169503
- [Background] George LK, Blazer DG, Hughes DC, Fowler N. Social support and the outcome of major depression. Br J Psychiatry. 1989 Apr;154:478-85. doi: 10.1192/bjp.154.4.478. PMID 2590779
- [Background] Green BH, Copeland JR, Dewey ME, Sharma V, Saunders PA, Davidson IA, Sullivan C, McWilliam C. Risk factors for depression in elderly people: a prospective study. Acta Psychiatr Scand. 1992 Sep;86(3):213-7. doi: 10.1111/j.1600-0447.1992.tb03254.x. PMID 1414415
- [Background] Hagan R, Manktelow R, Taylor BJ, Mallett J. Reducing loneliness amongst older people: a systematic search and narrative review. Aging Ment Health. 2014;18(6):683-93. doi: 10.1080/13607863.2013.875122. Epub 2014 Jan 17. PMID 24437736
- [Background] Hanson BS. Social network, social support and heavy drinking in elderly men--a population study of men born in 1914, Malmo, Sweden. Addiction. 1994 Jun;89(6):725-32. doi: 10.1111/j.1360-0443.1994.tb00958.x. PMID 8069173
- [Background] Heinrich LM, Gullone E. The clinical significance of loneliness: a literature review. Clin Psychol Rev. 2006 Oct;26(6):695-718. doi: 10.1016/j.cpr.2006.04.002. Epub 2006 Jun 19. PMID 16952717
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] House JS. Social isolation kills, but how and why? Psychosom Med. 2001 Mar-Apr;63(2):273-4. doi: 10.1097/00006842-200103000-00011. No abstract available. PMID 11292275
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Jessen F, Amariglio RE, van Boxtel M, Breteler M, Ceccaldi M, Chetelat G, Dubois B, Dufouil C, Ellis KA, van der Flier WM, Glodzik L, van Harten AC, de Leon MJ, McHugh P, Mielke MM, Molinuevo JL, Mosconi L, Osorio RS, Perrotin A, Petersen RC, Rabin LA, Rami L, Reisberg B, Rentz DM, Sachdev PS, de la Sayette V, Saykin AJ, Scheltens P, Shulman MB, Slavin MJ, Sperling RA, Stewart R, Uspenskaya O, Vellas B, Visser PJ, Wagner M; Subjective Cognitive Decline Initiative (SCD-I) Working Group. A conceptual framework for research on subjective cognitive decline in preclinical Alzheimer's disease. Alzheimers Dement. 2014 Nov;10(6):844-52. doi: 10.1016/j.jalz.2014.01.001. Epub 2014 May 3. PMID 24798886
- [Background] Kramarow EA. The elderly who live alone in the United States: historical perspectives on household change. Demography. 1995 Aug;32(3):335-52. PMID 8829970
- [Background] Luanaigh CO, Lawlor BA. Loneliness and the health of older people. Int J Geriatr Psychiatry. 2008 Dec;23(12):1213-21. doi: 10.1002/gps.2054. PMID 18537197
- [Background] Locher JL, Ritchie CS, Roth DL, Baker PS, Bodner EV, Allman RM. Social isolation, support, and capital and nutritional risk in an older sample: ethnic and gender differences. Soc Sci Med. 2005 Feb;60(4):747-61. doi: 10.1016/j.socscimed.2004.06.023. PMID 15571893
- [Background] Capron DW, Schmidt NB. Development and randomized trial evaluation of a novel computer-delivered anxiety sensitivity intervention. Behav Res Ther. 2016 Jun;81:47-55. doi: 10.1016/j.brat.2016.04.001. Epub 2016 Apr 8. PMID 27101256
- [Background] Masi CM, Chen HY, Hawkley LC, Cacioppo JT. A meta-analysis of interventions to reduce loneliness. Pers Soc Psychol Rev. 2011 Aug;15(3):219-66. doi: 10.1177/1088868310377394. Epub 2010 Aug 17. PMID 20716644
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Norr AM, Gibby BA, Schmidt NB. Is computerized psychoeducation sufficient to reduce anxiety sensitivity in an at-risk sample?: A randomized trial. J Affect Disord. 2017 Apr 1;212:48-55. doi: 10.1016/j.jad.2017.01.032. Epub 2017 Jan 23. PMID 28142083
- [Background] Ong AD, Uchino BN, Wethington E. Loneliness and Health in Older Adults: A Mini-Review and Synthesis. Gerontology. 2016;62(4):443-9. doi: 10.1159/000441651. Epub 2015 Nov 6. PMID 26539997
- [Background] O'Rourke HM, Collins L, Sidani S. Interventions to address social connectedness and loneliness for older adults: a scoping review. BMC Geriatr. 2018 Sep 15;18(1):214. doi: 10.1186/s12877-018-0897-x. PMID 30219034
- [Background] Piersol CV, Canton K, Connor SE, Giller I, Lipman S, Sager S. Effectiveness of Interventions for Caregivers of People With Alzheimer's Disease and Related Major Neurocognitive Disorders: A Systematic Review. Am J Occup Ther. 2017 Sep/Oct;71(5):7105180020p1-7105180020p10. doi: 10.5014/ajot.2017.027581. PMID 28809652
- [Background] Pressman SD, Cohen S, Miller GE, Barkin A, Rabin BS, Treanor JJ. Loneliness, social network size, and immune response to influenza vaccination in college freshmen. Health Psychol. 2005 May;24(3):297-306. doi: 10.1037/0278-6133.24.3.297. PMID 15898866
- [Background] Reeve BB, Hays RD, Bjorner JB, Cook KF, Crane PK, Teresi JA, Thissen D, Revicki DA, Weiss DJ, Hambleton RK, Liu H, Gershon R, Reise SP, Lai JS, Cella D; PROMIS Cooperative Group. Psychometric evaluation and calibration of health-related quality of life item banks: plans for the Patient-Reported Outcomes Measurement Information System (PROMIS). Med Care. 2007 May;45(5 Suppl 1):S22-31. doi: 10.1097/01.mlr.0000250483.85507.04. PMID 17443115
- [Background] Rico-Uribe LA, Caballero FF, Martin-Maria N, Cabello M, Ayuso-Mateos JL, Miret M. Association of loneliness with all-cause mortality: A meta-analysis. PLoS One. 2018 Jan 4;13(1):e0190033. doi: 10.1371/journal.pone.0190033. eCollection 2018. PMID 29300743
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Schmidt NB, Eggleston AM, Woolaway-Bickel K, Fitzpatrick KK, Vasey MW, Richey JA. Anxiety Sensitivity Amelioration Training (ASAT): a longitudinal primary prevention program targeting cognitive vulnerability. J Anxiety Disord. 2007;21(3):302-19. doi: 10.1016/j.janxdis.2006.06.002. Epub 2006 Aug 4. PMID 16889931
- [Background] Schmidt NB, Capron DW, Raines AM, Allan NP. Randomized clinical trial evaluating the efficacy of a brief intervention targeting anxiety sensitivity cognitive concerns. J Consult Clin Psychol. 2014 Dec;82(6):1023-33. doi: 10.1037/a0036651. Epub 2014 May 12. PMID 24821096
- [Background] Schmidt NB, Raines AM, Allan NP, Zvolensky MJ. Anxiety sensitivity risk reduction in smokers: A randomized control trial examining effects on panic. Behav Res Ther. 2016 Feb;77:138-46. doi: 10.1016/j.brat.2015.12.011. Epub 2015 Dec 21. PMID 26752327
- [Background] Schmidt NB, Norr AM, Allan NP, Raines AM, Capron DW. A randomized clinical trial targeting anxiety sensitivity for patients with suicidal ideation. J Consult Clin Psychol. 2017 Jun;85(6):596-610. doi: 10.1037/ccp0000195. Epub 2017 Mar 13. PMID 28287798
- [Background] Short NA, Stentz L, Raines AM, Boffa JW, Schmidt NB. Intervening on Thwarted Belongingness and Perceived Burdensomeness to Reduce Suicidality Among Veterans: Subanalyses From a Randomized Controlled Trial. Behav Ther. 2019 Sep;50(5):886-897. doi: 10.1016/j.beth.2019.01.004. Epub 2019 Jan 24. PMID 31422845
- [Background] Short NA, Boffa JW, King S, Albanese BJ, Allan NP, Schmidt NB. A randomized clinical trial examining the effects of an anxiety sensitivity intervention on insomnia symptoms: Replication and extension. Behav Res Ther. 2017 Dec;99:108-116. doi: 10.1016/j.brat.2017.09.013. Epub 2017 Oct 5. PMID 29035703
- [Background] Schumaker JF, Shea JD, Monfries MM, Groth-Marnat G. Loneliness and life satisfaction in Japan and Australia. J Psychol. 1993 Jan;127(1):65-71. doi: 10.1080/00223980.1993.9915543. PMID 8510053
- [Background] Short NA, Boffa JW, Norr AM, Albanese BJ, Allan NP, Schmidt NB. Randomized Clinical Trial Investigating the Effects of an Anxiety Sensitivity Intervention on Posttraumatic Stress Symptoms: A Replication and Extension. J Trauma Stress. 2017 Jun;30(3):296-303. doi: 10.1002/jts.22194. Epub 2017 Jun 6. PMID 28585746
- [Background] Short NA, Fuller K, Norr AM, Schmidt NB. Acceptability of a brief computerized intervention targeting anxiety sensitivity. Cogn Behav Ther. 2017 Apr;46(3):250-264. doi: 10.1080/16506073.2016.1232748. Epub 2016 Oct 7. PMID 27712458
- [Background] Silva C, Ribeiro JD, Joiner TE. Mental disorders and thwarted belongingness, perceived burdensomeness, and acquired capability for suicide. Psychiatry Res. 2015 Mar 30;226(1):316-27. doi: 10.1016/j.psychres.2015.01.008. Epub 2015 Jan 15. PMID 25650048
- [Background] Smith TF, Hirdes JP. Predicting social isolation among geriatric psychiatry patients. Int Psychogeriatr. 2009 Feb;21(1):50-9. doi: 10.1017/S1041610208007850. Epub 2008 Oct 30. PMID 18959811
- [Background] Stek ML, Vinkers DJ, Gussekloo J, Beekman AT, van der Mast RC, Westendorp RG. Is depression in old age fatal only when people feel lonely? Am J Psychiatry. 2005 Jan;162(1):178-80. doi: 10.1176/appi.ajp.162.1.178. PMID 15625218
- [Background] Steptoe A, Owen N, Kunz-Ebrecht SR, Brydon L. Loneliness and neuroendocrine, cardiovascular, and inflammatory stress responses in middle-aged men and women. Psychoneuroendocrinology. 2004 Jun;29(5):593-611. doi: 10.1016/S0306-4530(03)00086-6. PMID 15041083
- [Background] Stravynski A, Boyer R. Loneliness in relation to suicide ideation and parasuicide: a population-wide study. Suicide Life Threat Behav. 2001 Spring;31(1):32-40. doi: 10.1521/suli.31.1.32.21312. PMID 11326767
- [Background] Taylor SE, Repetti RL, Seeman T. Health psychology: what is an unhealthy environment and how does it get under the skin? Annu Rev Psychol. 1997;48:411-47. doi: 10.1146/annurev.psych.48.1.411. PMID 9046565
- [Background] Taylor HO, Taylor RJ, Nguyen AW, Chatters L. Social Isolation, Depression, and Psychological Distress Among Older Adults. J Aging Health. 2018 Feb;30(2):229-246. doi: 10.1177/0898264316673511. Epub 2016 Oct 17. PMID 28553785
- [Background] Thoits PA. Stress, coping, and social support processes: where are we? What next? J Health Soc Behav. 1995;Spec No:53-79. PMID 7560850
- [Background] Tilvis RS, Kahonen-Vare MH, Jolkkonen J, Valvanne J, Pitkala KH, Strandberg TE. Predictors of cognitive decline and mortality of aged people over a 10-year period. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):268-74. doi: 10.1093/gerona/59.3.m268. PMID 15031312
- [Background] Uchino BN. Social support and health: a review of physiological processes potentially underlying links to disease outcomes. J Behav Med. 2006 Aug;29(4):377-87. doi: 10.1007/s10865-006-9056-5. Epub 2006 Jun 7. PMID 16758315
- [Background] Van Orden KA, Witte TK, Gordon KH, Bender TW, Joiner TE Jr. Suicidal desire and the capability for suicide: tests of the interpersonal-psychological theory of suicidal behavior among adults. J Consult Clin Psychol. 2008 Feb;76(1):72-83. doi: 10.1037/0022-006X.76.1.72. PMID 18229985
- [Background] Van Orden KA, Cukrowicz KC, Witte TK, Joiner TE. Thwarted belongingness and perceived burdensomeness: construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychol Assess. 2012 Mar;24(1):197-215. doi: 10.1037/a0025358. Epub 2011 Sep 19. PMID 21928908
- [Background] Wang HX, Karp A, Winblad B, Fratiglioni L. Late-life engagement in social and leisure activities is associated with a decreased risk of dementia: a longitudinal study from the Kungsholmen project. Am J Epidemiol. 2002 Jun 15;155(12):1081-7. doi: 10.1093/aje/155.12.1081. PMID 12048221
- [Background] Wilson RS, Krueger KR, Arnold SE, Schneider JA, Kelly JF, Barnes LL, Tang Y, Bennett DA. Loneliness and risk of Alzheimer disease. Arch Gen Psychiatry. 2007 Feb;64(2):234-40. doi: 10.1001/archpsyc.64.2.234. PMID 17283291
- [Background] Yang YC, Boen C, Gerken K, Li T, Schorpp K, Harris KM. Social relationships and physiological determinants of longevity across the human life span. Proc Natl Acad Sci U S A. 2016 Jan 19;113(3):578-83. doi: 10.1073/pnas.1511085112. Epub 2016 Jan 4. PMID 26729882
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Berkman LF, Syme SL. Social networks, host resistance, and mortality: a nine-year follow-up study of Alameda County residents. Am J Epidemiol. 1979 Feb;109(2):186-204. doi: 10.1093/oxfordjournals.aje.a112674. PMID 425958